CLINICAL TRIAL: NCT06338982
Title: Fracture Pattern Following Bilateral Sagittal Split Osteotomy With or Without Impacted Third A Randomized Controlled Trial Assessing Fracture Pattern, Condylar Segment Positioning, Complications and Patient-reported Outcome Measures
Brief Title: Fracture Pattern Following Bilateral Sagittal Split Osteotomy With or Without Impacted Third Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kimie Bols Østergaard (Other)
Responsible Party: Sponsor-Investigator, Kimie Bols Østergaard, Doctor of Dental Surgery, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N-20230059
Record Dates: First submitted 2024-03-02; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Impacted Third Molar Tooth; Osteotomy; Orthognathic Surgery; Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures | interventions — beta-sitosterol oleate

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with a test group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group with interoperative wisdom tooth removal in conjunction with BSSO (Experimental)
  Interventions: Procedure: Interoperative wisdom tooth removal in conjunction with BSSO
- Control group with wisdom tooth removal at least 6 months before BSSO (No Intervention)

INTERVENTIONS:
Procedure: Interoperative wisdom tooth removal in conjunction with BSSO — The objective of the present randomized controlled trial is to assess the fracture pattern, condylar segment positioning, frequency of complications, and PROMs following BSSO with or without impacted mandibular third molars. this is illustrated by the fact that the test group had their wisdom teeth removed in connection with the sagittal split of the mandible (the BSSO surgery). Subsequently, all outcome measures are compared with the control group, who had their wisdom teeth removed 6 months prior their BSSO surgery.
  Arms: Test group with interoperative wisdom tooth removal in conjunction with BSSO

SUMMARY:
The goal of this clinical trial is to investigate the hypothesis that there are none difference in the treatment result of orthognathic surgery on the lower jaw, with interoperative wisdom tooth removal rather than preoperative wisdom tooth removal. In patients with severe dental malocclusion combined with a dentofacial deformity. The main question it aims to answer are:

• Is there a difference in the degree of complication and the patient's perception, with inter-operative wisdom tooth removal rather than pre-operative wisdom tooth removal.

Participants will be will be divided into two groups, with one group having their wisdom teeth removed 6 months before their jaw moving surgery and the other group having their wisdom teeth removed in connection with their jaw moving surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgical correction of facial deformities involving BSSO or bimaxillary surgery with bilateral asymptomatic impacted mandibular third molars
* Age between 18 and 75 years

Exclusion Criteria:

* Fully erupted and well-functioning mandibular third molar
* Unilateral impacted mandibular third molar
* Pathology associated with the impacted mandibular third molar
* BSSO combined with genioplasty
* Previous mandibular fractures
* Present neurosensory disturbances of the inferior alveolar nerve
* Systemic bone disease or arthritis
* Physical status classification system, ASA Class III or IV, specified patients with severe systemic disease ore patients with severe systemic disease that is constant threat to life
* Failure to attend the entire observation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Fracture pattern following BSSO with or without impacted third molars | 1 week after det BSSO surgery
  The fracture pattern of the mandible following BSSO will be assessed by CBCT scans (i-CAT; Imaging Sciences International, Hatfield, PA, USA) obtained preoperatively, and one week after surgery. The CBCT will be taken by fixed exposure parameters of 120 kV, 160 × 60 mm field of view, 0.30 mm voxel size, and 8.9-second images. The fracture pattern of the mandible will be classified according to LSS by the study investigator (KBØ). The LSS consisted of 4 categories based on the path of the fracture line on the lingual side of the mandibular ramus.
Condylar segment position following BSSO with or without impacted third molars | 1 week after det BSSO surgery
  The mandibular condylar segment positioning will be assessed in the sagittal, vertical, and transverse dimension by superimposing the pre- and postoperative CBCT scan using dedicated software (OnDemand3D Application, version 10; Cybermed, Seoul, South Korea). The orbital bony walls on the preoperative CBCT will be used as the reference and matched with the orbital walls on the postoperative CBCT. Pair-wise registration will be done, based on the automated detection of hundreds of virtual landmarks in the volumes, which can subsequently be manually adjusted, based on visible anatomical landmarks.To estimate the condylar displacement in all three dimensions, the intertransverse distance in millimeters between the center of the condyles is measured on the pre- and postoperative CBCT. Moreover, the distance between the mandibular condyle to the glenoid fossa is measured in the sagittal and vertical dimension. The measurements will be conducted by the study investigator (KBØ).
Oral Health Impact Profile-14 (OHIP-14) | Hand out questionnaires at the following five times, Enrolment, immediately prior to BSSO, One week after BSSO, One months after BSSO and One-year after BSSO
  OHIP-14 is a validated questionnaire for assessment of OHRQoL. OHIP-14 states the patient's overall oral impairment and does not take a specific treatment site into account. OHIP-14 is organized into seven conceptual dimensions including functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability and handicap. The response format of OHIP-14 is: Very often = 4; Fairly often or many times = 3; Occasionally = 2; Hardly ever or nearly never = 1; Never/I don´t know = 0. Thus, OHIP-14 scale ranged from 0 to 56 and dimension score ranged from 0 to 8. Values of the 14 items and each dimension are summed to calculate the OHIP-14 severity score and higher scores indicate poorer OHRQoL
The Modified Dental Anxiety Scale (MDAS) | Hand out questionnaires at the following three times, Enrolment, immediately prior to BSSO and One-year after BSSO
  The level of preoperative dental anxiety is assessed by MDAS, which is a brief questionnaire rating patient's emotional reaction to an up-coming dental visit.MDAS consist of five questions in a Likert scale ranging from not anxious (scoring 1), slightly anxious (scoring 2), fairly anxious (scoring 3), very anxious (scoring 4) to extremely anxious (scoring 5) and summed together to produce a total score ranging from 5 to 25. For assessing the level of dental anxiety of each patient, response scores of all 5 questions are added. The total score ranges from 5 to 25 with cut-off scores 14 and 19 suggestive of high dental anxiety and dental phobia.
Short Form-36 (SF-36) | Hand out questionnaires at the following five times, Enrolment, immediately prior to BSSO, One week after BSSO, One months after BSSO and One-year after BSSO
  SF-36 is a questionnaire for assessment of quality of life. SF-36 is composed of eight multi-item scales (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health), with scores for each of these scales (or dimensions) ranging from 0 to 100. Higher scores indicate higher health-related quality of life.
PROMs | Hand out questionnaires at the following two times, One week after BSSO and One months after BSSO.
  Patient´s perception of recovery will be assessed by questionnaires and visual analog scale ranging from 0 to 100 higher scores indicate bigger impact on the topic, the questions will assessing pain, number of days with sick leave, social and working isolation, physical appearance, eating and speaking ability, diet variations, sleep impairment, and discomfort as well as questions whether they would undergo similar treatment again, if needed or if they would recommend this treatment to a friend or a relative, if indicated.

SECONDARY OUTCOMES:
Length of the surgical procedure | Interoperative in connection with the BSSO surgery
  The intraoperative length of BSSO will be measured by a stopwatch (iPhone 14 Pro or similar) from the incision to the last suture in both groups. The intraoperative length of BSSO will be registered by the surgeon.
Intraoperative bleeding | Interoperative in connection with the BSSO surgery
  The intraoperative blood loss will be estimated by measuring suctioned blood, and then adjusted for the used volume of saline irrigation during BSSO. If the patient is undergoing bimaxillary surgery, then the blood loss will solely be calculated and registered for the BSSO. The intraoperative blood loss will be registered by the surgeon.
Frequency of intra- and postoperative complications | One week, one months and one-year after BSSO
  Frequency of intra- and postoperative complications including visualization and injury of the inferior alveolar nerve, heavy bleeding, or unfavorable fracture patterns will be registered by the surgeon.
  Postoperative complications including temporary or permanent neurosensory disturbances of the inferior alveolar nerve and infection will be registered by the surgeon. Infection will be registered according to the criteria for surgical site infection event (SSI) stated by the center of disease control.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg universitets hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No